CLINICAL TRIAL: NCT00369408
Title: Targeted Naltrexone for Problem Drinkers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Henry R. Kranzler, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 03-107-2; NIAAA-KRA-P50-03510
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-06

CONDITIONS: Alcoholism; Alcohol Drinking; Alcohol Dependence
Keywords: Randomized Trial; Medication for Heavy Drinking; Naltrexone Treatment; Daily vs. Targeted Administration
MeSH Terms: conditions — Alcoholism; Alcohol Drinking | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): naltrexone (50 mg orally) for 12-week treatment period
  Interventions: Drug: Naltrexone
- 2 (Placebo Comparator): placebo for 12-week treatment period
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Naltrexone — naltrexone (50 mg orally) for 12-week treatment period; 3 and 6 months post-treatment follow-up
  Other Names: ReVia
  Arms: 1
Drug: placebo — placebo for 12-week treatment period; 3 and 6 months post-treatment follow-up
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether naltrexone, combined with brief coping skills therapy, is effective in the treatment of heavy drinking.

DETAILED DESCRIPTION:
This is a 12-week, placebo-controlled trial of naltrexone (50 mg orally) in 163 problem drinkers. Problem drinkers are those individuals whose drinking puts them at risk of a variety of psychosocial and medical problems, including alcohol dependence, but who are not physically dependent on alcohol. They are estimated to comprise up to 20% of the general population. The study employed a factorial design in which the effects of medication (naltrexone vs. placebo), schedule of medication administration (i.e., daily vs. targeted), and the interaction of these factors on drinking behavior were examined. Targeted administration refers to the use of medication to cope with anticipated high-risk drinking situations.

The daily monitoring using interactive voice response technology of mood, desire to drink, perceived self-efficacy, and drinking behavior will make it possible to examine in depth the processes by which the study variables exert their effects. Daily monitoring was performed using automated telephone interviews, with in-person follow-up evaluations conducted at 3 and 6 months post-treatment to provide a measure of the durability of treatment effects.

A pharmacogenetic analysis based on preliminary evidence showing that a functional polymorphism in the gene encoding the mu-opioid receptor (OPRM1) affects response to naltrexone will serve to explore an important source of variation in the response to naltrexone treatment. Exploratory analyses involving other potential genetic moderators of the response to naltrexone, such as the gene encoding the delta opioid receptor (OPRD1), will also be conducted, as will the correlation of genotype data with other phenotypes.

Careful evaluation of the study hypotheses will provide important information on the efficacy and mechanism of the effects of targeted naltrexone in problem drinkers. This study will allow us to model effects across multiple levels of analysis in an effort to understand the psychopharmacological mechanisms underlying the therapeutic effects of naltrexone in problem drinkers and to apply novel genetic findings to understanding the pharmacogenetic mechanisms underlying the therapeutic effects of naltrexone in problem drinkers.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients 18-70 years of age.
* Participants will have an average weekly ethanol consumption of >=24 standard drinks for men, or >=18 standard drinks for women (i.e., substantially in excess of non-hazardous drinking levels).
* Participants will be able to read English at the eighth grade or higher level and show no evidence of significant cognitive impairment.
* If a woman of child-bearing potential (i.e., who has not had a hysterectomy, bilateral oophorectomy, tubal ligation or who are less than two years postmenopausal), participant must be non-lactating, practicing a reliable method of birth control, and have a negative serum pregnancy test prior to initiation of treatment.
* Participants will be willing to provide signed, informed consent to participate in the study (including a willingness to reduce drinking to non-hazardous levels).

Exclusion Criteria:

* Participants who have a current, clinically significant physical disease or abnormality on the basis of medical history, physical examination, or routine laboratory evaluation, including total bilirubin elevations of >110% or ALT or AST elevations >300% the upper limit of normal or have a diagnosis of Hepatitis B or C infection or AIDS (given the potential for adverse effects of naltrexone on liver function).
* Participants who have a serious psychiatric illness (i.e., schizophrenia, bipolar disorder, severe major depression, panic disorder, borderline personality states, organic mood or mental disorders, or substantial suicide or violence risk) on the basis of history or psychiatric examination.
* Participants who have a current Diagnostic and Statistical Manual of Mental Disorders 4th ed (DSM-IV) diagnosis of drug dependence (other than nicotine dependence) or a lifetime DSM-IV diagnosis of opioid dependence.
* Participants who have a current DSM-IV diagnosis of alcohol dependence that is clinically severe.
* Participants who have used opioids or other psychoactive medications regularly in the month prior to study enrollment.
* Participants who have a history of hypersensitivity to naltrexone.
* Participants who are considered by the investigators to be an unsuitable candidate for receipt of an investigational drug.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2003-06; Primary Completion 2007-08 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Drinking days and heavy drinking days | 12-week trial; 3 and 6 months post-treatment follow-up

SECONDARY OUTCOMES:
Alcohol-related problems | 12-week trial; 3 and 6 months post-treatment follow-up
Biological measures of alcohol consumption (i.e., serum GGTP and CDT) | 12-week trial; 3 and 6 months post-treatment follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Henry R. Kranzler, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

REFERENCES:
- [Result] Kranzler HR, Tennen H, Armeli S, Chan G, Covault J, Arias A, Oncken C. Targeted naltrexone for problem drinkers. J Clin Psychopharmacol. 2009 Aug;29(4):350-7. doi: 10.1097/JCP.0b013e3181ac5213. PMID 19593174